CLINICAL TRIAL: NCT07180628
Title: Organization and Development of Motor Cortical Circuits for Speech Production in Stuttering
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Soo-Eun Chang, Associate Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00269390; 1R01DC022763-01 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Stutter; Stuttering, Adult; Stuttering; Stuttering, Developmental
Keywords: Magnetic Resonance Imaging (MRI) scans; Behavioral assessments
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Intervention Model Description: There will be 50 adults that stutter that participate in this study with a goal of 33 evaluable.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stutter group (Experimental): Participants that stutter
  Interventions: Behavioral: Speech Production During functional magnetic resonance imaging (MRI)

INTERVENTIONS:
Behavioral: Speech Production During functional magnetic resonance imaging (MRI) — Participants will complete a speech production task with 2 conditions (stuttered, non-stuttered) while undergoing functional MRI to assess brain activity. Brain activity will be compared within subjects for the 2 conditions. The intervention is the combination of tasks delivered to all participants. The speaking task is the intervention (modifying agent) and the MRI is a measurement tool, not a therapeutic or modifying agent.

SUMMARY:
The overall objective of this study is to examine inter effector areas (IEAs) activity and functional connectivity during continuous speech production in stuttering adults.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18-65 years
* Have otherwise normal speech, language, hearing and cognition
* Speak English as their primary language
* Currently stutter

Exclusion Criteria:

* Have serious medical or neurological conditions (e.g., stroke, traumatic brain injury, Parkinson's disease, etc.)
* Have had a closed head injury (e.g., concussion)
* Have a reading disorder (e.g., dyslexia)
* Have hearing loss
* Have metal or electronic implants (e.g., cochlear implants, pacemakers, etc.)
* Are currently pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Blood-Oxygen-Level-Dependent (BOLD) signal change during speaking | During the speech task (5 runs, 8 minutes each) distributed across MRI Visits 1-6, up to 12 months from enrollment.
  The Blood-oxygen-level-dependent (BOLD) signal reflects changes in blood oxygenation levels that are associated with neural activity. It is measured using functional magnetic resonance imaging (fMRI) and reported in arbitrary units (a.u.). The BOLD response provides an indirect index of localized brain activity during task performance, with increased signal indicating greater activation in a given brain region relative to baseline or a comparison condition. In this study, BOLD signal differences will be compared within participants across two speech production tasks: (1) stuttered speech and (2) non-stuttered speech. Each participant will complete the speech task on several of the MRI visits, which varies per participant (total amount of time spent will be the same across participants).

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Eun Shang, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No